CLINICAL TRIAL: NCT00208286
Title: Clinical Evaluation of the P.F.C. Sigma (Fixed Bearing) and P.F.C. Sigma Rotating Platform (Mobile Bearing) Total Knee Systems.
Brief Title: P.F.C. Sigma Fixed Versus P.F.C. RP Mobile Bearing Total Knee Systems
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary study outcome achieved; investigator decided to conduct the study without sponsor support after 2009.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT0101
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PFC Sigma Fixed Bearing (Other): PFC Sigma Fixed Bearing system for use in total knee arthroplasty
  Interventions: Device: PFC Sigma Fixed Bearing
- PFC Sigma Mobile Bearing (Active Comparator): PFC Sigma Mobile Bearing system for use in total knee arthroplasty
  Interventions: Device: PFC Sigma Mobile Bearing

INTERVENTIONS:
Device: PFC Sigma Fixed Bearing — PFC Sigma Fixed Bearing system for use in total knee arthroplasty
  Arms: PFC Sigma Fixed Bearing
Device: PFC Sigma Mobile Bearing — PFC Sigma Mobile Bearing system for use in total knee arthroplasty
  Arms: PFC Sigma Mobile Bearing

SUMMARY:
This post-market clinical follow-up study was designed to compile long-term knee replacement outcomes of the PFC Sigma fixed and PFC Sigma mobile Rotating Platform (RP) knee systems. The first patient had surgery on November 8, 2001 and the final patient had surgery on July 29, 2005. There were 120 knees consented by a single site, which was the planned sample size in the study protocol, with 117 receiving one of the study devices. The study was terminated as the primary outcome was met and the investigator decided to conduct the study without sponsor support after 2009.

DETAILED DESCRIPTION:
Performance and safety will be assessed using the following surgeon and patient based outcome tools:

1. American Knee Society Knee and Function Scores
2. Knee Society Radiological Analysis
3. Oxford Knee Score
4. SF 12 Score
5. Anterior Knee Pain Score

Specific objectives of the evaluation being to assess the following:

1. Improvement in functional recovery
2. Incidence of anterior knee pain
3. Improvement in Quality of life
4. Incidence of tibial loosening
5. Incidence of excessive polyethylene wear

ELIGIBILITY:
Inclusion Criteria:

1. Administrative - The patient or their authorised representative is able to understand the evaluation, is able to give voluntary written informed consent and will comply with the post operative follow up regime.
2. Age - There are no restrictions relating to age of the patient. The patient's age must be considered suitable by the clinical investigator for a bi-compartmental or tri-compartmental knee arthroplasty using either of the two systems available in the evaluation.
3. Sex - Male or female (providing that they are not pregnant) may be recruited to the evaluation.
4. Diagnosis - patients that require a tri-compartmental knee arthroplasty for primary surgical management of idiopathic osteoarthritis.
5. Suitability - Patients who in the opinion of the Clinical Investigator are considered to be suitable for treatment with a fixed or mobile bearing tibial knee system and are suitable for patella resurfacing.

Exclusion Criteria:

1. Patients with rheumatoid arthritis.
2. Patients requiring revision total knee arthroplasty surgery.
3. Patients with any tibial deformity requiring tibial component augmentation.
4. Patients that in the opinion of the clinical investigators require a constrained prosthesis.
5. Patients with a known history of poor compliance to medical treatment.
6. Patients who are known drug or alcohol abusers.
7. Patients with a pathology which in the opinion of the clinical investigator will adversely affect healing.
8. Patients who are currently participating in another clinical evaluation.
9. Patients with other disorders which in the opinion of the Clinical Investigator will / could impair rehabilitation.
10. Contra-indications for use of the device, as detailed in the package insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-11; Primary Completion 2006-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To Compare Range of Motion (ROM) between subjects receiving Sigma Rotating Platform mobile bearing and Sigma fixed bearing components | 1 year
  Range of motion is knee flexion (how far the patient can bend their knee) minus knee extension (how far the patient can straighten their knee). The result of this subtraction is the range of motion (bending and straightening) for that knee.

SECONDARY OUTCOMES:
Change in SF-12 Physical and Mental Component Scores from Baseline to 1 and 2 years | 1 and 2 years
  The 12-Item Short Form Health Survey (SF-12) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-12) and Mental Component Score (MCS-12). At times, the survey is also displayed via 8 domain scales that are also scored from 0 to 100 (where 100 indicates the highest level of health) as follows: Physical Function, Role Physical, Bodily Pain, General Health, Mental Health, Role Emotional, Social Function, and Vitality. The response metric is the change score, or delta, from pre-operative assessment to post-operative assessment.
Change in American Knee Society Knee and Function Scores from Baseline to 1 and 2 years | 1 and 2 years
  American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability. American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee. The function score is composed of Walking and Stair Climbing ability.
Change in Oxford Knee Score from Baseline to 1 and 2 years | 1 and 2 years
  The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Change in Anterior Knee Pain from Baseline to 1 and 2 years | 1 and 2 years
  Anterior Knee Pain is assessed by the patient into 1 of 4 categories: None, Mild, Moderate, or Severe.
Incidence of Femoral Radiolucencies at one year | 6 weeks to 3 Months through 1 year
  Radiolucent lines (RLL) are looked for radiographically by component, from an AP view, and, if present and > 2mm, the number of knees is displayed.
Incidence of Tibial Radiolucencies at one year | 6 weeks to 3 Months through 1 year
  Radiolucent lines (RLL) are looked for radiographically by component, from an AP view, and, if present and > 2mm, the number of knees is displayed.
Incidence of Patellar Radiolucencies at one year | 6 weeks to 3 Months through 1 year
  Radiolucent lines (RLL) are looked for radiographically by component, from an AP view, and, if present and > 2mm, the number of knees is displayed.

CONTACTS AND LOCATIONS:
Locations (1):
- Middlesborough General Hospital, Middlesbrough, United Kingdom